CLINICAL TRIAL: NCT01315587
Title: A Double-blind Placebo Controlled Trial the Comparison of Effectiveness of Repetitive TMS and iTBS on Negative Symptoms and Cognition in Patients With Schizophrenia
Brief Title: Repetitive Transcranial Magnetic Stimulation and Intermittent Theta Burst (iTBS) in Schizophrenia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Tehran (Other)
Responsible Party: Principal Investigator, reza kazemi, Researcher, University of Tehran
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 23456
Record Dates: First submitted 2011-03-14; First posted 2011-03-15 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- intermittent theta burst stimulation (Active Comparator)
  Interventions: Device: repetitive Transcranial Magnetic Stimulation (Magstim rapid2 )
- repetitive Transcranial Magnetic Stimulation (Active Comparator)
  Interventions: Device: repetitive Transcranial Magnetic Stimulation (Magstim rapid2)
- Sham TMS (Placebo Comparator)
  Interventions: Device: repetitive Transcranial Magnetic Stimulation(Magstim rapid2)

INTERVENTIONS:
Device: repetitive Transcranial Magnetic Stimulation (Magstim rapid2 ) — * 3 pulses at 50Hz repeated each 200 ms for 2 seconds
  * 80% MT
  * 20 days treatment
  Other Names: TMS; rTMS; TBS; iTBS
  Arms: intermittent theta burst stimulation
Device: repetitive Transcranial Magnetic Stimulation (Magstim rapid2) — LDLPFC 110% MT 15 Hz 20 days
  Other Names: TMS; rTMS
  Arms: repetitive Transcranial Magnetic Stimulation
Device: repetitive Transcranial Magnetic Stimulation(Magstim rapid2) — Placebo treatment: Sham coil
  Arms: Sham TMS

SUMMARY:
The pilot studies have showed that theta burst stimulation (TBS) can have the more rapid and durable effects to the apply traditional rTMS protocols. The aim of this study is to investigate the effect of repetitive TMS and theta burst in reduction of negative symptoms and remission of cognitive functioning in patients with schizophrenia. In a randomized, double blind clinical trials, 30 patients with schizophrenia in Razi psychiatric hospital will be assigned to receive repetitive TMS; theta burst, or sham TMS, daily; for 20 sessions. The negative symptoms and cognitive functioning will be assessed before the treatment (pre test) during the treatment (session 10), and after the treatment (post test).QEEG and LORETA apply before and after rTMS in all subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients male and female with the range of 18-50 years of age
2. The diagnosis of schizophrenia according to DSM-IV-TR
3. Completion of consent form
4. Being under supervision of a psychiatrist,
5. Being able to adhere to treatment schedule,
6. Having stable symptoms as defined by not requiring a change in antipsychotic medication for at least 4 weeks or at least 2 weeks for psychotropic agents prior to entering the Study

Exclusion Criteria:

1. The history of rTMS treatment for any reason
2. Cardiac pacemaker
3. Drug pumps
4. Acute heart attack
5. The risk of seizure with any reasons
6. The history of epilepsy or seizure in the first relatives
7. Any metal in head
8. Brain trauma
9. Pregnancy
10. Breastfeeding
11. Drug dependency

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-01; Primary Completion 2015-11 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Positive and negative syndrome scale ( PANSS ) | Change of baseline in negative symptoms at 20 sessions

SECONDARY OUTCOMES:
Calgary depression for schizophrenia scale (CDSS) | 3 times (Before treatment, session 10, immediately after treatment)
  The CDSS is administered for measuring of depression before treatment, session 10, immediately after treatment
Schizophrenia quality of life scale (SQLS) | 3 times (Before treatment, session 10, immediately after treatment)
  The SQLS is administered for apprising of quality of life before treatment, session 10, immediately after treatment.
Cantab Schizophrenia Battery | 3 times (Before treatment, session 10, immediately after treatment)
  Cantab Schizophrenia Battery is included six tests, which is measuring for cognitive function. The cognitive function includes reaction time, executive function, Sustained attention, , Episodic memory . These scales:
  Reaction time (RTI) Rapid Visual information processing (RVP) Spatial Working Memory (SWM) One Touch Stockings of Cambridge (OTS) Paired Associates Learning (PAL) Intra-Extra Dimensional set- Shift (IED)
QEEG and low resolution brain electromagnetic tomography (LORETA) | 3 times (Before treatment,session 10, immediately after treatment)
  QEEG and LORETA is applying for assessment brain waves patterns.

OTHER OUTCOMES:
Hamilton Depression Rating Scale (HAMD-17) | 3 times (Before treatment,session 10, immediately after treatment)

CONTACTS AND LOCATIONS:
Locations (1):
- Atieh Clinical Neuroscience Center (ACNC), Tehran, Tehran Province, Iran